CLINICAL TRIAL: NCT01062529
Title: Peripheral Metabolic Effects of Intra Arterial Somatostatin Infusion in Healthy Controls
Brief Title: Peripheral Metabolic Effects of Somatostatin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: M-2008005
Record Dates: First submitted 2010-01-28; First posted 2010-02-04 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Acromegaly; Growth Hormone Deficiency; Diabetes
Keywords: GH signalling; insulin resistance; somatostatin; acromegaly
MeSH Terms: conditions — Acromegaly; Dwarfism, Pituitary; Diabetes Mellitus; Insulin Resistance | interventions — Somatostatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- somatostatin (Experimental)
  Interventions: Drug: Somatostatin

INTERVENTIONS:
Drug: Somatostatin — 4 h of 150 microgram infusion

SUMMARY:
The aim of this study is to investigate peripheral effects of Somatostatin on glucose metabolism and growth hormone (GH) signalling in healthy men. Eight subjects will be enrolled. The hypothesis is that Somatostatin infusion reverses insulin resistance caused by GH.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 27 kg/m2
* Written informed consent
* Healthy

Exclusion Criteria:

* Any disease
* Any use of medications
* Present or previous malignancy
* Alcohol dependency
* Allergy to trial medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Plasma levels of glucose | 3 months

SECONDARY OUTCOMES:
GH signalling | one year
Serum levels of free fatty acids (FFA) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, Professor, Principal Investigator
Locations (1):
- Medical department M, Aarhus, Aarhus, Denmark